CLINICAL TRIAL: NCT00139165
Title: Long-Term Treatment of Collagenous Colitis With Budesonide. Prospective, Doubleblind Placebo-Controlled Trial.
Brief Title: Long-Term Treatment of Collagenous Colitis With Budesonide
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bonderup, Ole K., M.D. (Individual)
Collaborators: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: okbon123
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2005-08

CONDITIONS: Collagenous Colitis
Keywords: Collagenous colitis; Budesonide treatment; Diarrhea
MeSH Terms: conditions — Colitis, Collagenous; Diarrhea | interventions — Budesonide; Sigmoidoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Budesonide — Capsule. Oral 6 mg o.d. for 24 weeks
Procedure: sigmoidoscopy — Sigmoidoscopy performed 2 times during the study period.

SUMMARY:
The aim of the trial is to examine the effect of budesonide treatment on collagenous colitis. All patients is treated for 6 weeks with budesonide and thereafter randomised to 24 weeks treatment with placebo or continued budesonide. The end poit is effect on clinical symptoms (number of daily stools)

ELIGIBILITY:
Inclusion Criteria:

* Histological criteria of Collagenous colitis
* Clinical activity (> 3 stools/day)

Exclusion Criteria:

* Treatment of Collagenous colitis within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2004-09; Study Completion 2006-03

PRIMARY OUTCOMES:
Clinical symptoms

SECONDARY OUTCOMES:
Histological changes

CONTACTS AND LOCATIONS:
Overall Officials: Ole K Bonderup, MD, Principal Investigator
Locations (2):
- Denmark (2):
  - Dept. of medical gastroenterology, Aalborg
  - Dept. of medical gastroenterology, Aarhus